CLINICAL TRIAL: NCT05395143
Title: Study to Assess the Effect of Zinc in Atorvastatin Treated Hyperlipidemic Patients: a Randomized, Double-blind, Placebo-controlled Trial
Brief Title: Study to Assess the Effect of Zinc in Atorvastatin Treated Hyperlipidemic Patients
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Bangabandhu Sheikh Mujib Medical University, Dhaka, Bangladesh (Other)
Responsible Party: Principal Investigator, Rumana Sharmin, principal investigator, Bangabandhu Sheikh Mujib Medical University, Dhaka, Bangladesh
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: BSMMU/2021/4030
Record Dates: First submitted 2022-05-24; First posted 2022-05-27 (Actual); Last update posted 2022-05-27 (Actual); Status verified 2022-05

CONDITIONS: Hyperlipidemias
Keywords: Atorvastatin; Zinc; Hyperlipidemia
MeSH Terms: conditions — Hyperlipidemias | interventions — Zinc Sulfate

STUDY DESIGN:
Intervention Model Description: A randomized, double-blind, placebo-controlled trial where one group consists of 46 hyperlipidemic patients under treatment with atorvastatin and zinc; and another group consists of 46 hyperlipidemic patients under treatment with atorvastatin and placebo
Who Masked: Participant, Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Atorvastatin and zinc (Experimental): 46 Hyperlipidemic patients are included in this arm who will receive Atorvastatin and Zinc. Zinc tablets of 30mg will be used once daily according to randomization along with Atorvastatin.
  Interventions: Drug: Zinc sulfate
- Atorvastatin and placebo (Placebo Comparator): 46 Hyperlipidemic patients are included in this arm who will receive Atorvastatin and placebo. Placebo tablets of 30mg will be used once daily according to randomization along with Atorvastatin.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Zinc sulfate — Zinc sulfate tablet 30mg once daily orally for 8 weeks along with Atorvastatin.
  Arms: Atorvastatin and zinc
Drug: Placebo — Placebo tablet 30mg once daily orally for 8 weeks along with Atorvastatin.
  Arms: Atorvastatin and placebo

SUMMARY:
This study was 8 weeks randomized, double-blind, placebo-controlled trial to assess the effect of zinc in Atorvastatin treated hyperlipidemic 92 patients. Participants were assessed at baseline, and 8 weeks. Subjects were randomized to receive either atorvastatin+placebo in one arm or atorvastatin +zinc 30mg tablet in another arm daily for 8 weeks. The outcome was the measure of fasting lipid profile, sgpt, serum creatinine at baseline and after 8 weeks following the intervention.

DETAILED DESCRIPTION:
Hyperlipidemia is a pathological disorder that includes raised concentration of serum cholesterol, LDL and triglycerides (TGs). It is one of the most important triggering factors for the development of cardiovascular disease. As a consequence, this disorder ultimately increases the mortality rate since cardiovascular disease (CVD) is globally the most common cause of death. Various studies have demonstrated that the prevalence rate of CVD in Bangladesh is 0.33% to 19.6% (Malik, A., 1976 and Zaman, M.M. et al, 2007) and hyperlipidaemia is 46%. Triglycerides, cholesterol, and lipoproteins are associated with the pathogenesis of coronary artery disease, especially atherosclerosis. Atherosclerotic lesions may be the consequence of reduced serum high-density lipoprotein (HDL) and increased triglycerides level. Triglyceride concentrations of about 1.7 mmol/L would be considered by many to be the point beyond which risk for coronary artery disease begins. Triglyceride concentrations are commonly increased in diabetes mellitus, particularly the insulin-resistant type, noninsulin-dependent diabetes mellitus (NIDDM), and indicate an enhanced risk of coronary artery disease. Hypercholesterolemia also enhances microvascular dysfunction by stimulating nitro-oxidative stress and induction of inflammation. This mechanism leads to the development of myocardial infarction. Normalization of serum lipid profile is the logical step to prevent atherosclerotic events such as myocardial infarction, ischaemic stroke, peripheral vascular disease and this will reduce the mortality rate. As hyperlipidemia is a flexible condition, it can be modified by alteration of dietary habit, lifestyle change, and applications of various medications which interfere with lipid metabolism with the body. In that case, statin medication is the most suitable therapy for hyperlipidemia. The 2014 ACC (American College of Cardiology) / AHA (American Heart Association) guidelines have highlighted the benefits of statin therapy. But despite the statins being very effective drug recommended target lipid lowering levels are not always achieved. Moreover, long-term high-dose statin therapy may give rise to some adverse effects. On the other hand, many other lipid lowering agents are available in the market but they are not able to achieve the target lipid lowering effect always and long term use of these drugs may promote some adverse effects. They are also costly. Therefore, exploration of alternative, affordable, efficacious with less adverse effects drugs should be the next point of interest for further study. Besides, the repeated incidence of cardiovascular disease brings lingering hazards for the health. This situation develops the requirement for an add-on lipid-lowering agent along with conventional statin therapy. In that case, Zinc could be an agent added along with conventional statin therapy to normalize the lipid profile. Zinc is an important micronutrient of the human body which is implicated as a component in various systemic wellbeing. Several studies found that zinc might have protective effect in the prevention of atherosclerosis. Effect of Zinc on lipid profile by some studies revealed that it can lower serum total cholesterol, LDL cholesterol, triglycerides and increase the HDL levels. Therefore, the current study will explore the combination of lipid-lowering activity of atorvastatin and zinc. This study will be a randomized, double blind, placebo controlled trial. It will be conducted in the department of pharmacology, BSMMU in collaboration with the department of cardiology, BSMMU.A total of 92 patients suffering from hyperlipidemia will be selected according to inclusion and exclusion criteria. The diagnosis of patients and the selection of drug and dosage would be performed by a senior professor of the cardiology department. After completing the necessary formalities including informed consent of the patients, they will be enrolled and randomly allocated into two arms: control arm and intervention arm. Patient in intervention arm would consist of 46 patients who will receive Atorvastatin plus Zinc (30 mg) tablet once daily orally for 8 weeks. On the other hand, control arm would consist of 46 patients who will receive Atorvastatin plus placebo for 8 weeks. The lipid profile will be measured at baseline and 8 weeks follow up

ELIGIBILITY:
Inclusion Criteria:

* Age: 18 to 75 years
* Sex: both male and female
* Hyperlipidemic patients suffering from ischemic heart disease, diabetes mellitus, hypertension.
* A person can develop hyperlipidemia if they have one or a combination of the following: Diagnostic criteria for dyslipidemic patients (NCEP ATP III guideline) Total Cholesterol > 240 mg/dl LDL-C > 100 mg/dl Triglyceride > 150 mg/dl HDL-C < 40 mg/dl

Exclusion Criteria:

* Patients with renal impairment.
* Patient with history of active liver disease (e.g. jaundice, hepatitis, cirrhosis)
* Patients having hypersensitivity to drugs.
* Patients with any systemic diseases or having serious infections or terminal illness (e.g.-tuberculosis, HIV, malignant tumor)
* Pregnant woman
* lactating mother

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 92 (Estimated)
Dates: Start 2021-05-01 (Actual); Primary Completion 2022-07-10 (Estimated); Study Completion 2022-07-10 (Estimated)

PRIMARY OUTCOMES:
Change of TC | from the baseline after 8-week treatment;

SECONDARY OUTCOMES:
Change of LDL-C | from the baseline after 8-week treatment
Change of HDL-C | from the baseline after 8-week treatment
Change of TG | from the baseline after 8-week treatment

CONTACTS AND LOCATIONS:
Locations (1):
- Bangabandhu Sheikh Mujib Medical University, Dhaka, Bangladesh